CLINICAL TRIAL: NCT02748005
Title: Asses the Efficacy of Furosap: A Testosterone Booster Supplement in Human Volunteers
Brief Title: Evaluation of Furosap in Human Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chemical Resources (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CR/TEST-5-14
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2015-08

CONDITIONS: Hypogonadism
Keywords: Fenugreek seed extract; testosterone; protodioscin; hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Furosap

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fenugreek seeds extract 500 mg (Experimental): Fenugreek seeds extract(Furosap) 500 mg
  Interventions: Dietary Supplement: Fenugreek seeds extract 500 mg

INTERVENTIONS:
Dietary Supplement: Fenugreek seeds extract 500 mg — one cap once a day
  Other Names: Furosap

SUMMARY:
The study evaluates the effect of Fenugreek seed extract (Furosap) in management of symptomatic hypogonadism as fenugreek seed extract is a testosterone booster. Fenugreek seeds extract are known to possess protodioscin and the extract is reported to improve sperm count, sperm morphology and protective effect on male reproductive system. All the participants will receive one capsule (500 mg) of furosap once a day.

DETAILED DESCRIPTION:
Testosterone deficiency (hypogonadism) is increasingly recognized as a significant health problem in aging men. Testosterone deficiency can adversely affect sexual function, physical health and psychological health. Consequently, the quality of life of men with low testosterone is negatively affected.

A certain proportion of middle-aged and elderly men have total testosterone concentrations below the reference range for young adult males. Possible consequences of reduced androgen levels include fat mass gain, loss of muscle and bone mass, fatigue, depression, anaemia, poor libido and erectile dysfunction. The clinical features of androgen deficiency in the aging male (ADAM) resemble those of hypogonadism of younger subjects, with a single relevant difference: each of these features can also occur in elderly men with normal androgen levels.

The world Health Organization estimates that by 2025, worldwide, the number of people aged over 65 years will rise from the current figure of 390 million to 800 million. In the Hypogonadism in Males (HIM) study of men treated in the primary care setting, 38.7% of men aged ≥45 years tested positive for hypogonadism (TT <300 ng/dL). Applied to U. S. census data, these findings suggest that 13.8 million American men aged ≥45 years may be testosterone- deficient. Furthermore, the prevalence of testosterone deficiency increases with age, reaching 50% for men aged ≥85 years. As the population ages, the burden of testosterone deficiency is expected to grow. The prevalence of low testosterone also increases in men with common co- morbidities, such as obesity, diabetes, and metabolic syndrome.

The nutritional status with an age is a major determinant of health and fitness. Nutrition plays a central role in adaptation, rehydration, refueling, and repair as well as recovery from injury and other problems. The testosterone supplementation in older men with low testosterone levels may improve the testosterone level which further improve the physical, sexual, and cognitive functions, and improve mood and quality of life FUROSAP® is an innovative product made through a novel patented process, involving physical separations of active ingredients from the seeds of Fenugreek herb (Trigonella foenum-graecum) without affecting chemical properties of the active fractions. It is a natural and promising dietary supplement. It"s dietary supplement comprising Protodioscin as the major fraction which isolated from fenugreek seeds.

Protodioscin is the active ingredient found in the extract of the plant. Protodioscin increases levels of the hormones testosterone, dihydrotestosterone and dehydroepiandrosterone. It boosts testosterone level via stimulating pituitary gland. Protodioscin acts by stimulating the enzyme 5- alpha-reductase, which plays a role in the conversion of testosterone into dihydrotestosterone. Dihydrotestosterone, in turn enhances erythropoiesis and muscle development. More erythropoiesis or production of red blood cell increases the haemoglobin level, which results in better oxygen transport throughout the body, resulting in a more optimal health. Both increased production of testosterone contribute to the increase in sexual functions, and it increases unbound free testosterone levels, which improves muscle mass, fat loss, strength and endurance. In addition, protodioscin also stimulates the hypothalamus secretion of luteinizing hormone (LH) which also helps to increase the level of testosterone.

ELIGIBILITY:
Inclusion Criteria:

1. Agrees to written as well as audio-visual informed consent.
2. Ability to understand the risks/benefits of the protocol
3. Male between 35-65 years of age.
4. Diagnosed with Symptomatic hypogonadism

Exclusion Criteria:

1. Uncooperative Subjects
2. Impaired hepatic function indicated by SGOT/SGPT >2.5 times the upper limit of normal.
3. Abnormal liver or kidney function tests (ALT or AST > 2 times the upper limit of normal
4. elevated creatinine, males > 125 µmol/L or 1.4mg/dl, females > 110 µmol/L or1.2mg/dl)
5. Patients suffering from CAD
6. History of malignancy
7. History of hypersensitivity to any of the investigational drugs Receiving any other testosterone booster therapy/medication/supplement within the last 2 months
8. History of coagulopathies
9. High alcohol intake (>2 standard drinks per day)
10. History of psychiatric disorder that may impair the ability of subjects to provide written informed consent.
11. Any medical condition, where the investigator feels participation in the study could be detrimental to the subjects overall well-being

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
% change in Serum Testosterone level | On completion of treatment (i.e.12 weeks) as compared to baseline
% improvement in sperm count | On completion of treatment (i.e.12 weeks) as compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Saroj Hospital & Maternity Centre, Kanpur Hardoi Ring Road, Para,Lucknow, U P, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steels E, Rao A, Vitetta L. Physiological aspects of male libido enhanced by standardized Trigonella foenum-graecum extract and mineral formulation. Phytother Res. 2011 Sep;25(9):1294-300. doi: 10.1002/ptr.3360. Epub 2011 Feb 10. PMID 21312304
- [Background] Aswar U, Bodhankar SL, Mohan V, Thakurdesai PA. Effect of furostanol glycosides from Trigonella foenum-graecum on the reproductive system of male albino rats. Phytother Res. 2010 Oct;24(10):1482-8. doi: 10.1002/ptr.3129. PMID 20878698
- [Background] Hamden K, Jaouadi B, Carreau S, Aouidet A, El-Fazaa S, Gharbi N, Elfeki A. Potential protective effect on key steroidogenesis and metabolic enzymes and sperm abnormalities by fenugreek steroids in testis and epididymis of surviving diabetic rats. Arch Physiol Biochem. 2010 Jul;116(3):146-55. doi: 10.3109/13813455.2010.486405. PMID 20507258
- [Background] Gauthaman K, Ganesan AP, Prasad RN. Sexual effects of puncturevine (Tribulus terrestris) extract (protodioscin): an evaluation using a rat model. J Altern Complement Med. 2003 Apr;9(2):257-65. doi: 10.1089/10755530360623374. PMID 12804079